CLINICAL TRIAL: NCT04944628
Title: An Observational Prospective Study to Evaluate the Efficacy of 2 Weeks of Oral Supplementation With a Probiotic Formula in Infants With Functional Gastrointestinal Disorders (FGDI)
Brief Title: Observational Prospective Study With Probiotic Supplementation on Infants With FGDI
Status: Completed | Type: Observational
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Other Study IDs: Normocolic ADL
Record Dates: First submitted 2021-06-14; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Functional Gastrointestinal Disorders; Infantile Colic; Functional Constipation
Keywords: FGDI; probiotic
MeSH Terms: conditions — Gastrointestinal Diseases; Colic | interventions — Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic in liquid format (oil suspension) administered 10 drops once daily for 2 weeks (2x10^9 cfu/day)

SUMMARY:
This observational prospective study evaluates the safety, tolerability and efficacy of a probiotic formula in infants with functional gastrointestinal disorders (FGDI)

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGDIs) affect one out of two infants during the fist six months of life and do not have an organic cause. Infant colic, so-called excessive crying syndrome, and functional constipation are among the most common paediatric FGDIs.

FGDIs pathophysiology is multifactorial and may include phycological factors and alterations of the gut physiology including gut microbiota dysbiosis.

Probiotics are proposed as a potential treatment for FGDIs. However, evidence is limited.

A probiotic formula composed of strains Bifidobacerium longum CECT 7894 and Pediococcus pentosaceus CECT 8330 is tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastrointestinal symptoms related to FGID including functional constipation and/or infant colic diagnosed according to Rome IV criteria for clinical purposes.
* ≥ 37 weeks of gestation at birth.
* ≥ 2500 g of birth weight.

Exclusion Criteria:

* Infants with failure to thrive (weight gain <100 grams/week on average from birth).
* Major medical problems (e. g. immunodeficiencies, developmental problems or genetic abnormalities)
* Gastrointestinal diseases
* Administered with antibiotics for 4 weeks or probiotics for 2 weeks before or during study

Ages: 1 Month to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population selected from primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Change in total FGDI severity | Day 1 and day 14
  FGDI severity measured as summatory of excessive crying score (5-point Likert scale (0: no symptoms, to 4: extremely severe symptoms) + constipation score (5-point Likert scales (0: no symptoms, to 4: extremely severe symptoms)

SECONDARY OUTCOMES:
Change in excessive crying severity | Day 1 and day 14
  Excessive crying score measured using 5-point Likert scales (0: no symptoms, to 4: extremely severe symptoms)
Change in constipation severity | Day 1 and day 14
  Constipation score measured using 5-point Likert scales (0: no symptoms, to 4: extremely severe symptoms)
Change in parental anxiety | Day 1 and day 14
  Recorded through the validated Generalized Anxiety Disorder (GAD) 7-item scale (GAD-7).
Tolerability and safety | Daily from day 1 to day 14
  Any adverse events experienced throughout study period
Parental satisfaction with the product | Day 14
  Measured with a 5-point Likert scale (0: very dissatisfied, to 4: very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Maura Sticco, MD, Principal Investigator — Azienda Sanitaria Locale Napoli
Locations (1):
- Azienda Sanitaria Locale Napoli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Derived] Asto E, Huedo P, Altadill T, Aguilo Garcia M, Sticco M, Perez M, Espadaler-Mazo J. Probiotic Properties of Bifidobacterium longum KABP042 and Pediococcus pentosaceus KABP041 Show Potential to Counteract Functional Gastrointestinal Disorders in an Observational Pilot Trial in Infants. Front Microbiol. 2022 Jan 12;12:741391. doi: 10.3389/fmicb.2021.741391. eCollection 2021. PMID 35095783